CLINICAL TRIAL: NCT04748614
Title: Comparative ICU Cost, Hospital Stay and Mortality Analysis Before and After COVID 19
Brief Title: Analysis Before and After COVID 19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Kocaeli Derince Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Merve Yazici Kara, MD, Kocaeli Derince Education and Research Hospital
Other Study IDs: Ilke-ICU
Record Dates: First submitted 2021-02-08; First posted 2021-02-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Cost of ICU
MeSH Terms: interventions — Costs and Cost Analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Before SARS-Cov2: Before SARS-Cov2
  Interventions: Other: Cost
- After SARS-Cov2: After SARS-Cov2
  Interventions: Other: Cost

INTERVENTIONS:
Other: Cost — ICU cost

SUMMARY:
In our study, we aimed to compare the average length of stay, death rates and costs of intensive care patients in October-November-December 2019 (before COVID 19) and October-November-December 2020 (during COVID 19).

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old
* All patients in intensive care unit in last three months of 2019
* All SARS-Cov2 patients in intensive care unit in last three months of 2020

Exclusion Criteria:

* Under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in intensive care in the last 3 months of 2019 and all SARS-Cov2 patients hospitalized in intensive care in the last 3 months of 2020.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Cost of ICU | 1 month
  Cost of ICU

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Khan AA, AlRuthia Y, Balkhi B, Alghadeer SM, Temsah MH, Althunayyan SM, Alsofayan YM. Erratum: Khan, A.A., et al. Survival and Estimation of Direct Medical Costs of Hospitalized COVID-19 Patients in the Kingdom of Saudi Arabia (Short Title: COVID-19 Survival and Cost in Saudi Arabia). Int. J. Environ. Res. Public Health 2020, 17, 7458. Int J Environ Res Public Health. 2020 Dec 17;17(24):9458. doi: 10.3390/ijerph17249458. PMID 33348933
- See also: WHO Coronavirus Disease (COVID-19) Dashboard — http://covid19.who.int/